CLINICAL TRIAL: NCT05167721
Title: Randomized Double-Blind Placebo-Controlled Adaptive Design Trial Of Intrathecally Administered Autologous Mesenchymal Stem Cells In Multiple System Atrophy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wolfgang Singer, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-005569; FD-R-07290-01 (Other: FDA OOPD)
Record Dates: First submitted 2021-11-30; First posted 2021-12-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple System Atrophy
Keywords: mesenchymal stem cells; treatment trial
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blind Placebo-Controlled Adaptive Design Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): 25 million mesenchymal stem cells administered intrathecally every 3 months for 4 injections
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- Arm 2 (Active Comparator): 25 million mesenchymal stem cells administered intrathecally every 6 months for 2 injections (placebo injections at 3 month and 9 month timepoints)
  Interventions: Biological: Autologous Mesenchymal Stem Cells; Other: Placebo
- Arm 3 (Placebo Comparator): Placebo (lactated Ringer's) administered intrathecally every 3 months for 4 injections
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells — Autologous Mesenchymal Stem Cells administered intrathecally
  Arms: Arm 1; Arm 2
Other: Placebo — Placebo administered intrathecally
  Arms: Arm 2; Arm 3

SUMMARY:
Multiple system atrophy (MSA) is a rare, rapidly progressive, and invariably fatal neurological condition characterized by autonomic failure, parkinsonism, and/or ataxia. There is no available treatment to slow or halt disease progression. The purpose of this study is to assess optimal dosing frequency, effectiveness and safety of adipose-derived autologous mesenchymal stem cells delivered into the spinal fluid of patients with MSA.

Funding source: FDA Office of Orphan Product Development (OOPD), Mayo Clinic Executive Dean for Research Transformational Award, Mayo Clinic Regenerative Medicine, and Mayo Clinic Department of Neurology.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a rare, rapidly progressive, and invariably fatal neurodegenerative disease for which there is no disease-modifying treatment. Recent insights into pathophysiologic mechanisms suggest a crucial role of deprivation of neurotrophic factors which have been shown to be secreted by mesenchymal stem cells (MSCs). In a recent phase I/II study adipose-derived autologous MSCs were delivered intrathecally to patients with early MSA utilizing a dose-escalation design. At a dose of 50 million MSCs, injections were generally well tolerated, but thickening of cauda equina nerve roots was observed which was either asymptomatic or associated with low back pain. The rate of disease progression assessed using the Unified MSA Rating Scale (UMSARS) was markedly slower compared to a matched control group. An even more favorable side effect profile and virtually lack of disease progression was seen in an add-on cohort receiving 25 million MSCs per injection. Neurofilament light chain, an index of central axonal degeneration, decreased in all patients receiving that dose. MSC administrations resulted in a marked, dose-dependent increase of neurotrophic factors in CSF. 2-year survival was significantly higher than observed in natural history cohorts.

Based on these findings we are now conducting a double-blind, placebo-controlled, adaptive design phase II trial of adipose-derived intrathecal autologous MSCs in MSA with the goal to establish optimal treatment frequency and simultaneously derive placebo-controlled efficacy and safety data in preparation for a multicenter phase III trial. Up to 76 adult subjects with MSA will be enrolled. To ensure a homogenous patient population with comparable rates of disease progression, we will restrict the study to early cases but still fulfilling strictest diagnostic consensus criteria. Participants will undergo a subcutaneous fat biopsy to derive autologous MSCs, which are cultured, expanded, and prepared for delivery in Mayo's Cell Therapeutics Lab. In a first phase, subjects will be randomized 1:1:1 to receive 25 million MSCs at two different injection intervals (every 6 months or every 3 months) as the two active arms or lactated Ringer's solution as the placebo arm. An interim analysis will take place after approximately 38 patients have completed the trial with assessments of the primary endpoint available at all timepoints. Additional patients enrolled after the first 38 patients and before the results of the interim analysis are available will receive the higher frequency administration utilizing 2:1 randomization. The DSMB will review efficacy and safety/tolerability data available at the time of the interim analysis and pick a "winner" based on efficacy trends and adverse events. The study will then continue utilizing 2:1 randomization ("winner" active: placebo). Patients undergo clinical assessments at baseline, 3, 6, 9, and 12 months to derive the primary endpoint, the rate of disease progression assessed using UMSARS total and a mixed effects regression model. MRI of the head and lumbar spine will be completed at baseline and 12 months to expand safety data and to assess the rate of atrophy of selected brain regions using morphometric measures as surrogate markers of disease progression. Spinal fluid before and after administrations, as well as stem cell product media will be collected to further explore biological properties and effects of MSCs and to assess selected spinal fluid markers as biomarkers of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 30-70 years, who are willing and able to give informed consent.
2. Clinical diagnosis of MSA, fulfilling consensus criteria for probable MSA.
3. UMSARS I (omitting question 11) between 5 and 17, and able to walk unaided (i.e. able to walk at least 50 yards without the use of a cane or walker, and without other support such as holding on to an arm or touching walls).
4. Anticipated survival of at least 3 years in the opinion of the investigator.
5. Normal cognition as assessed by the Montreal Cognitive Assessment (MOCA). We will require a value ≥26.

Exclusion Criteria:

1. Pregnant or breastfeeding women, and women of childbearing potential who do not agree to practice an acceptable method of birth control. Acceptable methods of birth control in this study are: surgical sterilization, intrauterine devices, partner's vasectomy, a double-protection method (condom or diaphragm with spermicide), hormonal contraceptive drug (i.e., oral contraceptive, contraceptive patch, long-acting injectable contraceptive) with a required second mode of contraception.
2. Participants with a clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the study or might affect study results. These include conditions causing significant CNS or autonomic dysfunction, clinically significant peripheral neuropathy, active malignant neoplasm, amyloidosis, active autoimmune disease, immunocompromised state, active infection, congestive heart failure (NYHA III or IV), recent (<6 months) myocardial infarction, history of stoke with residual deficits, uncontrolled diabetes mellitus, alcoholism, orthopedic problems that compromise mobility and activity of daily living, significant liver or kidney disease, thrombocytopenia (<50 x 109/L), disorders affecting coagulation, and patients on active anticoagulation.
3. Participants who have taken any investigational products within 90 days prior to baseline, or with expected effects lasting beyond 60 days prior to baseline.
4. Medications that could affect clinical evaluations are permitted but need to be withdrawn at least four half-lives prior to study visits. Those include medications used to treat motor symptoms, such as levodopa and other anti-Parkinsonian medications.
5. Patients with contraindication to any of the study procedures, in particular MRI scanning.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in UMSARS total (= UMSARS I + UMSARS II) score | 12 months
  Rate of disease progression assessed using the change in the UMSARS total (= UMSARS I + UMSARS II) score

SECONDARY OUTCOMES:
Change in UMSARS II score | 12 months
  Rate of disease progression assessed using the change in the UMSARS II subscore
Change in UMSARS I score | 12 months
  Rate of disease progression assessed using the change in the UMSARS I subscore
Change in modified UMSARS scale | 12 months
  Rate of disease progression assessed using a modified UMSARS scale comprising selected items of UMSARS that reflect clinically most meaningful aspects of the disease
Change in NfL | 9 - 12 months
  Change in NfL in CSF over time as biomarker of disease progression in MSA
Rate of atrophy of selected brain regions | 12 months
  Rate of atrophy of selected brain regions assessed using MRI morphometry (change from baseline to 12 months)
Change in COMPASS select score | 12 months
  Progression of autonomic symptoms assessed using COMPASS select

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Singer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials